CLINICAL TRIAL: NCT00175214
Title: Controlled Trial to Increase Detection and Treatment of Osteoporosis in Older Patients With a Wrist Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHFMR#2000000389
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Osteoporosis; Wrist Fractures
Keywords: osteoporosis; wrist fractures; quality improvement; knowledge translation
MeSH Terms: conditions — Osteoporosis; Wrist Fractures | interventions — Patient Education as Topic

INTERVENTIONS:
Behavioral: Multifaceted intervention (patient education, physician guidelines, reminders)

SUMMARY:
The primary objective of this proposed research is to improve the quality of care for patients who present to the Emergency Department with osteoporosis and a fracture of the wrist, by increasing the use of proven efficacious osteoporosis treatment. This is the primary study outcome, and it is defined as starting any one of hormone therapy, a bisphosphonate, raloxifene, or calcitonin within 6 months of a fracture of the wrist.

The study hypothesis is that a quality improvement intervention (with multiple components that include a notification system for primary care physicians, patient-specific reminders, locally generated treatment guidelines endorsed by opinion leaders, and patient education and counseling) will lead to increased use of proven efficacious osteoporosis treatments in patients eligible for secondary prevention. This hypothesis will be tested by comparing the intervention with usual care controls, in a prospective nonrandomized controlled trial.

DETAILED DESCRIPTION:
BACKGROUND: Osteoporosis is a progressive condition that causes a loss of bone mass, skeletal fragility, and fractures. Fractures result in pain, disability, deformity, and death. Osteoporosis is a major population health problem affecting 1.4 million Canadians, 25% of women and 12% of men over the age of 50 years. Current guidelines recommend aggressive secondary prevention in patients with osteoporosis who have suffered a fracture, because these patients have as high as a 20% risk of fracture in the following year, and because there are now proven efficacious treatments that can reduce this risk by 40-60%. Nevertheless, recent studies have shown that these patients are under-recognized and under-treated, demonstrating a care gap between evidence-based best practice and usual care. All patients with osteoporotic fractures (i.e., of the hip, vertebrae, or wrist) benefit from treatment. However, patients who present with a wrist fracture may be best suited to an intervention to improve secondary prevention practices, because wrist fractures are "sentinel events" in the natural history of osteoporosis: they are common, easily diagnosed, always present to medical attention, and occur years before the more devastating and costly fractures of the hip and vertebrae.

OBJECTIVES: The primary objective of this study is to improve the quality of care for patients who present to the ED with osteoporosis and a fracture of the wrist, by increasing the use of proven efficacious osteoporosis treatment. This is the primary study outcome, and it is defined as starting any one of hormone replacement therapy, a bisphosphonate, raloxifene, or calcitonin within 6 months of a fracture of the wrist.

HYPOTHESIS: A quality improvement intervention directed at patients and their primary care physicians will increase the use of proven efficacious osteoporosis treatment. The intervention itself has multiple components that include: a notification system and patient-specific reminders for primary care physicians, locally developed treatment guidelines endorsed by opinion leaders, and patient education and counseling. The study hypothesis will be tested by comparing the intervention to usual care controls, in a prospective nonrandomized controlled trial.

SPECIFIC AIMS: To determine whether the proposed intervention can-

* 1. Increase the use of proven efficacious osteoporosis treatment in patients with a fracture of the wrist,
* 2. Increase appropriate use of bone mineral density testing,
* 3. Increase patients' knowledge of osteoporosis and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years
* any closed distal forearm fracture
* discharged home

Exclusion Criteria:

* unwilling or unable to provide consent
* admitted to hospital
* long term care resident
* residence outside Edmonton, Alberta
* unable to read and converse in English
* currently taking prescription osteoporosis treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2001-01; Study Completion 2005-01

PRIMARY OUTCOMES:
Increased use of proven efficacious osteoporosis treatment within six months of study enrollment, defined as: hormone therapy, a bisphosphonate, raloxifene, or calcitonin.

SECONDARY OUTCOMES:
1. BMD testing
2. Osteoporosis diagnosis
3. Osteoporosis related knowledge
4. Satisfaction
5. Generic, Disease Specific, and Function-related QOL
6. Falls, falls-related injuries, and fall interventions
7. Persistence of effects and generalizability of effects
8. 1, 2, 3 year outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Sumit R Majumdar, MD, MPH, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospitals, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Majumdar SR, Rowe BH, Folk D, Johnson JA, Holroyd BH, Morrish DW, Maksymowych WP, Steiner IP, Harley CH, Wirzba BJ, Hanley DA, Blitz S, Russell AS. A controlled trial to increase detection and treatment of osteoporosis in older patients with a wrist fracture. Ann Intern Med. 2004 Sep 7;141(5):366-73. doi: 10.7326/0003-4819-141-5-200409070-00011. PMID 15353428
- [Derived] Majumdar SR, Johnson JA, Lier DA, Russell AS, Hanley DA, Blitz S, Steiner IP, Maksymowych WP, Morrish DW, Holroyd BR, Rowe BH. Persistence, reproducibility, and cost-effectiveness of an intervention to improve the quality of osteoporosis care after a fracture of the wrist: results of a controlled trial. Osteoporos Int. 2007 Mar;18(3):261-70. doi: 10.1007/s00198-006-0248-1. Epub 2006 Nov 4. PMID 17086470